CLINICAL TRIAL: NCT03285048
Title: Cognitive Remediation Therapy (CRT) for Adults Treated for Cancer: A Single-arm Proof of Concept Study.
Brief Title: Cognitive Remediation Therapy (CRT) for Adults Treated for Cancer
Acronym: CaCRT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MIRB 02072 MB0018
Record Dates: First submitted 2017-01-10; First posted 2017-09-15 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2018-10

CONDITIONS: Cancer of the Prostate; Cancer
Keywords: cognitive impairment
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasms; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cognitive Remediation Therapy (Experimental): Cognitive Remediation Training is comprised of 8 weeks of active cognitive training using Brain HQ auditory and visual training tasks. Training is twice per week for up to 2 hours. Also included is a Bridging Group at each training session. The Bridging group provides information about cognitive training and compensatory strategies to generalize the benefits of training to daily life.
  Interventions: Behavioral: Cognitive Remediation Therapy

INTERVENTIONS:
Behavioral: Cognitive Remediation Therapy — Brain HQ is a computer based cognitive training that uses hierarchical adaptive technology to provide challenging and demanding training that is not too frustrating or discouraging. Training includes auditory and visual sensory training, memory and executive function exercises. The Bridging group is based on similar training programs that focus on self-regulation training, problem focused cognitive behavior therapy and compensatory cognitive strategies.
  Other Names: Cognitive Remediation Training

SUMMARY:
This study is to determine the safety, feasibility and acceptability of an 8-week cognitive remediation training (CRT) in patients treated for cancer. The secondary objective of the study is to estimate the effect size of CRT in improving neurocognitive functioning and quality of life. This is a single-arm proof of concept study. Patients treated for cancer with persistent cognitive complaints will be recruited from the outpatient clinic of the VA Comprehensive Cancer Center, West Haven, CT, Yale Medicine, and greater New Haven community.The active treatment phase will be followed by an assessment at the conclusion of treatment to evaluate changes in cognitive function and quality of life. Participants will be invited back to participate in a final follow-up assessment 2 months later.

DETAILED DESCRIPTION:
Objectives:

The primary objective of this study is to determine the safety, feasibility and acceptability of an 8-week cognitive training intervention in patients treated for cancer. The secondary objective of the study is to estimate the effect size of CRT in improving neurocognitive functioning and quality of life for three different populations of cancer patients.

Research Design:

This is a single-arm proof of concept study with three cancer groups. Patients treated for cancer with persistent cognitive complaints will be recruited from the outpatient clinic of the VA Comprehensive Cancer Center, West Haven, CT, Yale Medicine, and greater New Haven community. We intend to enroll approximately 30 participants, with approximately 10 from each of the following cancer treatment types (1) participants who are at least six months from completion of adjuvant chemotherapy or chemoradiation and are in remission; (2) participants who are receiving long-term chemotherapy (6 months or longer) with a diagnosis of Stage IV cancer and with stable medical condition; (3) participants who are receiving long-term (6 months or longer) hormone therapy (androgen deprivation therapy or anti-estrogen therapy). Patients in this group who received chemotherapy will be eligible if they completed chemotherapy at least 6 months prior to enrolling. There will be an eight-week intervention period and a two-month follow-up assessment.

Methodology:

Participants will participate in a pre-assessment to establish eligibility, baseline cognitive function, and quality of life. This will be followed by participation in a cognitive remediation program (Brain HQ) for eight weeks during which all participants receive up to 16 hours of computerized cognitive training and 16 45-minute Bridging groups where they learn cognitive skills for daily living. The active treatment phase will be followed by an assessment at the conclusion of treatment to evaluate changes in cognitive function and quality of life. Participants will be invited back to participate in a final follow-up assessment 2 months later.

ELIGIBILITY:
Inclusion Criteria:

1.Participants who:

1. are at least six months from completion of adjuvant chemotherapy or chemoradiation and are in remission or;
2. are receiving long-term chemotherapy (6 months or longer) with a diagnosis of Stage IV cancer and with stable medical conditions or;
3. are receiving long-term (6 months or longer) hormone therapy (androgen deprivation therapy or anti-estrogen therapy). Patients in this group who received chemotherapy will be eligible if they completed chemotherapy at least 6 months prior to enrolling.

2. Subjective reports of cognitive decline. 3. Report that they are interested in seeking treatment to address their cognitive concerns.

4. Age 18 or older. 5. Fluency in English and a 6th grade or higher reading level.

Exclusion Criteria:

1. Does not meet one of the three participant categories
2. Unstable medical condition.
3. History of, or current symptoms of, serious psychiatric disorder requiring antipsychotic medications or hospitalization.
4. Current substance abuse disorder.
5. History of, or current central nervous system (CNS) malignancies, CNS radiation, intrathecal chemotherapy, or CNS-involved surgery.
6. Current IQ estimate less than 80.
7. Unable to give written informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01; Primary Completion 2017-08 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Self-report of daily cognitive function | 8 weeks
  Self-reported cognitive function includes symptoms of perceived cognitive impairments, perceived cognitive abilities, and overall quality of life. These are aggregated into a classification of overall degree of impairment and disability

SECONDARY OUTCOMES:
Neurocognitive function | 8 weeks
  Neurocognitive assessments using neurocognitive tests of attention, processing speed, executive function and memory changes from baseline. Results are aggregated into an overall score reflecting neurocognitive change from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Morris D Bell, Ph.D., Principal Investigator — Yale University
Locations (1):
- VA Connecticut Healthcare System, West Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No